CLINICAL TRIAL: NCT06673992
Title: Evaluation of Corneal Irregular Astigmatism and Visual Quality Following Bilateral Sequential Small Incision Lenticule Extraction (SMILE) and Laser Subepithelial Keratomileusis (LASEK): A Six-Year Comparative Study
Acronym: SMILE LASEK
Status: Completed | Type: Observational
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Hua Li, resident doctor, Shanghai 10th People's Hospital
Other Study IDs: Shanghai10HLi00001
Record Dates: First submitted 2024-10-26; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: This study does not involve any interventions — This study does not involve any interventions

SUMMARY:
To compare the corneal spherical component (SC), regular astigmatism (RA), irregular astigmatism (IA, including Asymmetry and Irregularity) and visual quality six years after small incision lenticule extraction (SMILE) and laser subepithelial keratomileusis (LASEK) for mild to moderate myopia.

ELIGIBILITY:
Inclusion Criteria:

* (1) patients aged over 18 years; (2) absence of corneal, ocular, or systemic diseases; (3) stable refractive diopter maintained for the past 2 years with a change of ± 0.50 diopter; (4) discontinuation of soft contact lens wear for at least 2 weeks and rigid contact lenses for at least 4 weeks prior to surgery; (5) preoperative manifest refraction spherical equivalent (MRSE) less than -6.00 diopter (D)

Exclusion Criteria:

A history of moderate to severe dry eye as well as any ocular or systemic disease that would contraindicate laser refractive surgery

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients with mild to moderate myopia or myopic astigmatism who underwent SMILE or LASEK between October 2017 and May 2018 were enrolled
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Corneal Irregular Astigmatism | preoperative and 6 years postoperatively
  The swept-source anterior segment OCT (CASIA SS-1000) was utilized to acquire corneal topography measurements. In the Corneal Map mode, 16 radial cross-sectional images (512 telecentric+A-scans) were obtained within a duration of 0.3 s for each measurement. The analysis program identified and digitized the anterior and posterior corneal surfaces to evaluate distributions of corneal power and corneal height for both the anterior and posterior corneal surfaces. The unit of Corneal Irregular Astigmatism is D.
wavefront aberration | preoperative and 6 years postoperatively
  The wavefront aberrations were measured and analyzed for 6-mm pupil diameter with a Zywave aberrometer using a Hartmann-Shack sensor (Bausch & Lomb, US). The absolute Zernike coefficients including vertical trefoil, horizontal trefoil, vertical coma, horizontal coma, spherical aberration, and total higher-order aberrations (tHOAs) were examined. The unit of wavefront aberration is um.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai 10th People's Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li H, Hu W, Li M, Shi Y, Sun L, Ma X, Zou J. Evaluation of Corneal Irregular Astigmatism and Visual Quality Following Bilateral Sequential SMILE and LASEK: A Six-Year Comparative Study. J Ophthalmol. 2026 Feb 8;2026:5989651. doi: 10.1155/joph/5989651. eCollection 2026. PMID 41669707